CLINICAL TRIAL: NCT03677297
Title: Comparative Evaluation of Treatment Of Infrabony Defects With and Without 1.2% Rosuvastatin Gel: In-Vivo Study
Brief Title: "Efficacy Of 1.2% Rosuvastatin Gel In The Management Of Infrabony Defects"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, DR. SUKHADA DEO, Principal investigator, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DPU/R & R (D)/ 98(10)/ 16
Record Dates: First submitted 2018-08-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Adult Periodontitis
Keywords: Intervention Study; Rosuvastatin; Periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ROSUVASTATIN (Experimental): 1.2% Rosuvastatin Gel. Insertion in infrabony defects once
  Interventions: Drug: Rosuvastatin
- placebo (Placebo Comparator): No intervention used on control site
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Test sites were treated with access flap surgery and 1.2% Rosuvastatin gel
  Other Names: No intervention used on Control site

SUMMARY:
Study aims to evaluate clinical and radiographic effectiveness of 1.2% Rosuvastatin gel in the treatment of Infrabony defects in chronic periodontitis patients.

DETAILED DESCRIPTION:
Source from where the patients will be selected:

10 patients with chronic periodontitis having two or more infrabony defects will be selected from the Outpatient section of Dept. of Periodontology, Dr. D. Y. Patil Dental College and Hospital, Pimpri, Pune - 18.

A detailed clinical examination, case history and written consent will be obtained from all the participants.

Before surgery, each patient will be given careful instructions regarding proper oral hygiene measures. A full-mouth phase I therapy will be performed. A periodontal re-evaluation will be performed after 4 to 6 weeks of phase 1 therapy to confirm the desired sites for the study. The selected sites will be divided randomly by using a Sequentially numbered, opaque, sealed envelopes (SNOSE) randomization into control and test sites. The control site will be treated with Access Flap Surgery (AFS), whereas test sites will be treated with AFS and 1.2% Rosuvastatin gel. Suitable antibiotics and analgesics will be prescribed along with Chlorhexidine digluconate rinses (0.2%) twice daily for 14 days. Patients will be examined at 4 weeks, 3 and 6 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 30-50 years
* Probing pocket depth ≥ 5mm following initial therapy.
* Suitable interproximal angular infrabony defects of ≥3mm.
* Involved teeth should be vital and asymptomatic.
* Systemically healthy patients.
* Patients who demonstrate acceptable oral hygiene prior to access flap surgery.
* Patients agreed to sign informed consent and willing to return for the follow up visits.

Exclusion Criteria:

* Systemic statin therapy
* Known or suspected allergy to the statin group
* Allergy to sulfur containing drugs
* History of aggressive periodontitis.
* Presence of gingival recession at the surgical site.
* Mobility of study teeth ≥ grade I.
* Use of tobacco in any form.
* Pregnant and lactating women.
* patients who have received any anti-inflammatory drugs and antibiotics in the previous six months.
* H/O osteoporosis.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Bone fill | 6 months
  Radiographic parameter measuring distance from cemento-enamel junction to the base of the defect.
  Difference in the measurement at the end of 6 months shows the amount of bone fill

SECONDARY OUTCOMES:
Probing depth | 6 months
  Clinical parameters- Reduction in this parameter is desired at the end of 6 months
relative attachment level | 6 months
  Clinical parameters- Reduction in this parameter at the end of 6 months shows gain in attachment
plaque index | 6 months
  Clinical parameters- Reduction in plaque index at the end of 6 months shows improvement in gingival health
bleeding index | 6 months
  Clinical parameters- Reduction in bleeding index at the end of 6 months shows improvement in gingival health

CONTACTS AND LOCATIONS:
Overall Officials: Sukhada D Deo, BDS, Principal Investigator — Dr. D. Y. Patil Dental College & Hospital
Locations (1):
- Sukhada Deo, Pune, Maharashtra, India